CLINICAL TRIAL: NCT06871241
Title: Public Awareness and Understanding of Palliative Care in the United Arab Emirates: Insights from a Population-Based Cross-Sectional Study
Brief Title: Public Awareness and Understanding of PC in the UAE
Status: Completed | Type: Observational
Sponsor: Burjeel Medical City (Other)
Responsible Party: Principal Investigator, Humaid O. Al-Shamsi, Chief Executive Officer, Burjeel Medical City
Organization: Burjeel Cancer Institute (Other)
Other Study IDs: BH/REC/073/24
Record Dates: First submitted 2025-02-03; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Palliative Care
Keywords: Supportive care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Palliative care (PC) is essential medical care for improving the quality of life for patients with life-threatening illnesses and their families. There has been substantial evolution of PC services in the United Arab Emirates (UAE), yet public awareness regarding PC remains shallow, hindering its utilization and acceptance on a large scale.

DETAILED DESCRIPTION:
This study aimed to evaluate public perceptions and awareness of PC in the UAE. A cross-sectional survey was conducted in both Arabic and English. This study emphasizes the need of addressing these gaps to integrate PC effectively into the UAE healthcare system, ensuring equitable access and improved quality of life for patients and their families.

ELIGIBILITY:
Inclusion Criteria:

* UAE residents
* Provided informed consent to participate
* Completed the survey in either Arabic or English

Exclusion Criteria:

* Non-UAE residents
* Incomplete survey responses (if applicable)

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The target population included residents of the UAE, both Emiratis and expatriates, who could read and respond in either English or Arabic.
Sampling Method: Non-Probability Sample
Enrollment: 824 (Actual)
Dates: Start 2024-07-25 (Actual); Primary Completion 2024-08-18 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Familiarity and Understanding of Palliative and Supportive Care as Measured by a Structured Survey | Surveys were conducted in Arabic from July 25, 2024, to August 18, 2024, and in English from August 5, 2024, to August 18, 2024.
  The study assessed participants' awareness, familiarity, and understanding of palliative and supportive care through a structured questionnaire. The survey includes Likert-scale and multiple-choice questions designed to evaluate:
  * Self-reported familiarity with palliative and supportive care concepts
  * Knowledge of available palliative care services
  * Perceived importance of palliative care in the healthcare system
  * Disparities in responses between Arabic-speaking and English-speaking groups.
  Responses were analyzed quantitatively by calculating the proportion of participants at different familiarity levels i.e., Very familiar, somewhat familiar, Neutral/not sure, not very familiar, not familiar at all and comparing trends across language groups. Percentages were calculated and categorical responses were summarized using frequency distributions.

CONTACTS AND LOCATIONS:
Locations (1):
- Burjeel Cancer Institute, Abu Dhabi, Abu Dhabi Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) from this study will not be publicly disclosed due to confidentiality concerns. However, aggregated data supporting the findings of this study may be available from the corresponding author upon reasonable request, subject to institutional and ethical approvals.